CLINICAL TRIAL: NCT03326024
Title: Long Term Assessment of Ovarian Reserve After More Than Two Years of Laparoscopic Ovarian Drilling in Polycystic Ovary Syndrome
Brief Title: The Ovarian Reserve and Laparoscopic Ovarian Drilling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Salama, Resident, Assiut University
Other Study IDs: 17100367
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- A: Patients with Polycystic Ovary Syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and underwent laparoscopic ovarian drilling from more than two years.
- B: Patients with Polycystic Ovary Syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and didn't undergo laparoscopic ovarian drilling

SUMMARY:
Long term assessment of ovarian reserve after more than two years of laparoscopic ovarian drilling in Polycystic Ovary Syndrome

DETAILED DESCRIPTION:
Inclusion criteria:

Goup "A": Patients with polycystic ovary syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and underwent laparoscopic ovarian drilling from more than two years.

Goup "B": Patients with polycystic ovary syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and didn't undergo laparoscopic ovarian drilling

Anti-mullerian hormone (as an indicator for ovarian reserve) will be measured for the two groups and data collected will be compared

ELIGIBILITY:
Inclusion Criteria:

* Goup "A": Patients with polycystic ovary syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and underwent laparoscopic ovarian drilling from more than two years.

Goup "B": Patients with polycystic ovary syndrome at reproductive age (20-35) diagnosed according to Rotterdam criteria and didn't undergo laparoscopic ovarian drilling

Exclusion Criteria:

1. Age <19 or > 35 years.
2. BMI <19 or > 35
3. patients refusing to participate in the study.
4. previous ovarian cystectomy.

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: OUPATIENT CLINICS OF women health hospital - Assiut university
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Level of anti-mullerian hormone after laparoscopic ovarian drilling | 2 years